CLINICAL TRIAL: NCT00002669
Title: TREATMENT OF METASTATIC MELANOMA WITH DTIC, CDDP AND IFN ALPHA WITH OR WITHOUT IL-2: A RANDOMIZED PHASE III TRIAL
Brief Title: Combination Chemotherapy, Interferon Alfa, and Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-18951; EORTC-18951
Record Dates: First submitted 2000-06-02; First posted 2003-04-11 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interferon-alpha; Cisplatin; Dacarbazine

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Drug: cisplatin
Drug: dacarbazine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of the cancer cells. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. It is not yet known which treatment regimen is more effective in treating melanoma.

PURPOSE: Randomized phase II trial to compare the effectiveness of two regimens of combination chemotherapy plus interferon alfa and interleukin-2 in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the rate of disease stabilization in patients with metastatic melanoma when treated with interferon alfa, dacarbazine, cisplatin, and interleukin-2.
* Assess toxicity, overall response rate, and response duration in these patients when treated with this regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive dacarbazine IV over 1 hour and cisplatin IV over 3 hours on days 1-3. Patients also receive interferon alfa subcutaneously (SQ) on days 1-5 and interleukin-2 by continuous IV infusion on days 4-9. Treatment continues every 28 days for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive dacarbazine IV on day 1 and 22 every 28 days for 2 courses. Patients then receive treatment as in arm I for a maximum of 4 courses.

Patients are followed every 2 months for 6 months, then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 42-90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma that is metastatic and unresectable
* Measurable, progressive disease (by physical exam and/or noninvasive imaging)

  * No prior irradiation of indicator lesions
* No CNS metastases (confirmed by CT or MRI)

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Greater than 3 months

Hematopoietic:

* WBC at least 2,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* No serious hepatic disease

Renal:

* Creatinine no greater than 1.65 mg/dL
* No serious renal disease

Cardiovascular:

* No serious cardiac disease

Pulmonary:

* No serious pulmonary disease

Other:

* No organ allograft
* No autoimmune disease
* No uncontrolled infection
* No active peptic ulcer
* No hyper or hypothyroidism
* No requirement for corticosteroids
* No second malignancy except basal cell skin carcinoma or carcinoma in situ of the cervix
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy with interleukin-2
* No prior interferon alfa in combination with cisplatin or dacarbazine

Chemotherapy:

* No prior chemotherapy with cisplatin in combination with dacarbazine
* More than 3 months since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 1995-06; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Study Chair — Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin
Locations (24):
- Landeskrankenanstalten - Salzburg, Salzburg, Austria
- Belgium (4):
  - Hopital Universitaire Erasme, Brussels
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- France (3):
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - Centre Leon Berard, Lyon
  - CHU Pitie-Salpetriere, Paris
- Germany (6):
  - Universitaetsklinikum Charite, Berlin
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Robert Roessle Klinik, Berlin
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Johannes Gutenberg University, Mainz
  - III Medizinische Klinik Mannheim, Mannheim
- Istituto Europeo Di Oncologia, Milan, Italy
- Netherlands (2):
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Instituto Portugues de Oncologia do Porto, Porto, Portugal
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitaetsspital, Zurich
- United Kingdom (4):
  - St. James's Hospital, Leeds, England
  - Royal Marsden NHS Trust, London, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - Royal Bournemouth Hospital, Bournemouth

REFERENCES:
- [Background] Agarwala SS, Keilholz U, Gilles E, Bedikian AY, Wu J, Kay R, Stein CA, Itri LM, Suciu S, Eggermont AM. LDH correlation with survival in advanced melanoma from two large, randomised trials (Oblimersen GM301 and EORTC 18951). Eur J Cancer. 2009 Jul;45(10):1807-14. doi: 10.1016/j.ejca.2009.04.016. Epub 2009 May 4. PMID 19419855
- [Background] Keilholz U, Suciu S, Bedikian AY, et al.: LDH is a prognostic factor in stage IV melanoma patients (pts) but is a predictive factor only for bcl2 antisense treatment efficacy: re-analysis of GM301 and EORTC18951 randomized trials. [Abstract] J Clin Oncol 25 (Suppl 18): A-8552, 485s, 2007.
- [Background] Keilholz U, Eggermont AM. The role of interleukin-2 in the management of stage IV melanoma: the EORTC melanoma cooperative group program. Cancer J Sci Am. 2000 Feb;6 Suppl 1:S99-103. PMID 10685668
- [Result] Schmidt H, Suciu S, Punt CJ, Gore M, Kruit W, Patel P, Lienard D, von der Maase H, Eggermont AM, Keilholz U; American Joint Committee on Cancer Stage IV Melanoma; EORTC 18951. Pretreatment levels of peripheral neutrophils and leukocytes as independent predictors of overall survival in patients with American Joint Committee on Cancer Stage IV Melanoma: results of the EORTC 18951 Biochemotherapy Trial. J Clin Oncol. 2007 Apr 20;25(12):1562-9. doi: 10.1200/JCO.2006.09.0274. PMID 17443000
- [Result] Punt CJ, Suciu S, Gore MA, Koller J, Kruit WH, Thomas J, Patel P, Lienard D, Eggermont AM, Keilholz U. Chemoimmunotherapy with dacarbazine, cisplatin, interferon-alpha2b and interleukin-2 versus two cycles of dacarbazine followed by chemoimmunotherapy in patients with metastatic melanoma: a randomised phase II study of the European Organization for Research and Treatment of Cancer Melanoma Group. Eur J Cancer. 2006 Nov;42(17):2991-5. doi: 10.1016/j.ejca.2006.08.012. Epub 2006 Oct 4. PMID 17023156
- [Result] Keilholz U, Punt CJ, Gore M, Kruit W, Patel P, Lienard D, Thomas J, Proebstle TM, Schmittel A, Schadendorf D, Velu T, Negrier S, Kleeberg U, Lehman F, Suciu S, Eggermont AM. Dacarbazine, cisplatin, and interferon-alfa-2b with or without interleukin-2 in metastatic melanoma: a randomized phase III trial (18951) of the European Organisation for Research and Treatment of Cancer Melanoma Group. J Clin Oncol. 2005 Sep 20;23(27):6747-55. doi: 10.1200/JCO.2005.03.202. PMID 16170182
- [Result] Keilholz U, Punt CJ, Gore M, et al.: Dacarbazine, cisplatin and interferon alpha with or without interleukin-2 in advanced melanoma: interim analysis of EORTC trial 18951. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A2043, 530a, 1999.